CLINICAL TRIAL: NCT07347210
Title: Evaluation of UCPVax Vaccine +/- Pembrolizumab Combined With Standard Treatment as Adjuvant Therapy in Patients With Unmethylated MGMT Glioblastoma: a Randomized Phase II Trial
Brief Title: Evaluation of UCPVax Vaccine +/- Pembrolizumab Combined With Standard Treatment as Adjuvant Therapy in Patients With Unmethylated MGMT Glioblastoma
Acronym: MATVAC-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/894; 2024-514399-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-21; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Primary Glioblastoma
Keywords: GBM; UCPVax; pembrolizumab; cancer vaccine; telomerase; CD4 T cell
MeSH Terms: interventions — pembrolizumab; Temozolomide

STUDY DESIGN:
Intervention Model Description: Randomization 2:2:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Arm A (Experimental): UCPVax + Pembrolizumab + Standard of care
  Interventions: Drug: UCPVax; Drug: Pembrolizumab; Drug: Temozolomide
- Experimental Arm B (Experimental): UCPVax + Standard of care
  Interventions: Drug: UCPVax; Drug: Temozolomide
- Control Arm C (Other): Standard of care
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: UCPVax — Priming : UCPVax (two helper peptides UCP2 and UCP4 + Montanide ISA51) at 0.5 mg subcutaneously at day 1, 8, 15, 29, 36 and 43
  Boost : UCPVax at 0.5 mg subcutaneously one month after priming and then every 8 weeks for 12 months maximum
  Arms: Experimental Arm A; Experimental Arm B
Drug: Pembrolizumab — 400 mg/m1 every 6 weeks since day 1 until disease progression or unacceptable toxicity for a maximum of 1 year
  Arms: Experimental Arm A
Drug: Temozolomide — 150-200 mg/m2/day x 5 days per month x 6 months according to best standard of care starting at day 1 of week 1 (with vaccine 1 of UCPVax).
  Additional treatment with NOVO-TTF200A will be allowed.

SUMMARY:
Glioblastomas (GBM) are the most frequent brain tumors and one of the most lethal adult cancers despite maximal multimodal therapy. Despite maximal safe resection followed by radiotherapy and temozolomide (TMZ) ± tumor-treating fields, median overall survival for newly diagnosed GBM remains around 18 months and long-term survival is rare, and recurrence is nearly universal. So, the development of new therapeutic strategies is a critical unmet need in GBM.

Despite the limited success of anti-PD(L)-1 therapy, immunotherapy remains a promising option in GBM. Current challenge supports to develop combinatorial therapy approaches considering the particular immune tumor microenvironment in GBM. Anticancer vaccines have shown promising signs of efficacy in GBM but critical factors challenge their efficacy. CD4 T help is of major interest for cancer vaccine effectiveness and for immune checkpoint inhibitors success. We previously designed UCPVax a CD4 T helper-targeted cancer vaccine derived from telomerase (TERT), a very attractive GBM-associated antigen (Adotévi O, J Clin Oncol 2023 ; Laheurte C, Cell Report Med 2025). The induction of robust tumor reactive CD4 T cell response with UCPVax together with TMZ-mediated immune effects will promote recruitment of effectors immune cells into tumor bed creating a more suitable microenvironment for anti-PD-1 action.

This is a proof-of-concept phase II trial to evaluate the efficacy of maintenance therapy evaluating UCPVax +/- pembrolizumab combined to standard treatment in newly diagnosed unmethylated MGMT glioblastoma. A translational research network will be implemented to better understand the therapeutic efficacy of this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 with informed consent signed
2. Patient with a confirmed histological diagnosis of non-mutated IDH primary glioblastoma (surgical resection or biopsy).
3. Tumor with unmethylated MGMT promoter status
4. Patients having completed the concomitant phase of radiotherapy + temozolomide regimen (standard radiotherapy with 60 Gy in 30 fractions or hypofractionated radiotherapy with 40 Gy in 15 fractions), and eligible for the 6 monthly cycles of maintenance temozolomide
5. Karnofsky Perfomance status (KPS) ≥ 70%
6. Life expectancy ≥ 3 months
7. If patient is treated by corticosteroïds (CS), patient must be on stable CS dose for 15 days and total daily dose ≤ 10 mg prednisone, or equivalent
8. Adequate organ function laboratory values
9. Females must be using highly effective contraceptive measures, and have a negative pregnancy test prior to the start of dosing if of childbearing potential, or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening :

   * Post-menopausal is defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
   * Women under the age of 50 years would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution.
   * Women with documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but tubal ligation.

   Female with childbearing potential must use effective contraception during study treatment and after the end of treatment based on the last study drug administrated: 6 months after the last dose of Temozolomide; 4 months after the last dose of pembrolizumab and 1 month after the last injection of UCPVax.
10. Male patients with a female partner of childbearing potential should be willing to use barrier contraception and to refrain from donating sperm during the study and and post-treatment based on the last study drug administrated: 3 months after the last dose of temozolomide; 4 months after the last pembrolizumab dose; 1 month after the last UCPVax injection.
11. Patient affiliated to or beneficiary of French social security system
12. Ability to comply with the study protocol, in the Investigator's judgment.
13. Signed and dates informed consent

Exclusion Criteria:

Patients will not be eligible for this study for any of the following reasons:

Cancer specific exclusion criteria:

1. IDH1 or IDH2 mutated tumor
2. Presence of extracranial metastasis
3. Leptomeningeal disease on MRI
4. Contrast enhancement ≥4 cm (largest diameter on axial T1 sequences) on inclusion MRI
5. Previous treatment with Carmustine impregnated wafers (GliadelR)
6. Previous treatment with bevacizumab or other Vascular Endothelial Growth Factor (VEGF) antagonists
7. Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study.

   Non-eligible to treatment by UCPVax:
8. Prior therapy with an anti-PD-1, anti-PD-L1, or with an agent directed to another immune checkpoint (e.g. CTLA-4, TIGIT, Lag3…).
9. Immunosuppressive treatment including CS > 10 mg prednisone or equivalent within the previous 2 weeks
10. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.
11. Has a known history of Human Immunodeficiency Virus (HIV) infection.
12. History of tuberculosis infection
13. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
14. Active auto-immune disease that has required a systemic treatment in the past 2 years (i.e. corticosteroïds or immunosuppressors). Replacement therapy (e.g. thyroxine, insulin) is allowed.
15. Active or history of auto-immune disease or immune deficiency
16. History of solid organ transplant nor allogenic hematopoietic stem cell transplantation
17. Hypersensitivity to the active substance temozolomide or to any of the excipients listed (anhydrous lactose, colloidal anhydrous silica, sodium carboxymethyl starch type A, tartaric acid, stearic acid),
18. Hypersensitivity to dacarbazine (DTIC)
19. Hypersensitivity to the active substance pembrolizumab or to any of the excipients listed (L-histidine, L-histidine hydrochloride monohydrate, sucrose, polysorbate 80 (E433))
20. Hypersensitivity to the active substance Montanide
21. Uncontrolled active systemic fungal, bacterial, viral, or other infection within the previous 4 weeks or requirement for intravenous (IV) antibiotics within the last two weeks
22. Inadequate hematology and organ functions; known cardiac failure or unstable coronaropathy, respiratory failure or another life threatening condition.
23. Patient with unresolved non-hematologic toxicities > Grade 1 (or > Grade 2 if deemed acceptable by the investigator and not considered a safety risk)
24. Major surgery within 1 month prior randomization or planned during the study
25. Vaccination with alive attenuated vaccine within 4 weeks prior the first dosing. Patient must agree not to receive live attenuated vaccine including influenza vaccine during the treatment and within 6 months following the last dose of pembrolizumab

    Non-eligible to a clinical trial:
26. Diagnosis of another malignant tumor within 2 years before randomization except treating resected basocellular carcinoma and carcinoma in situ such as breast cancer, endometrial or cervical carcinoma that have undergone curative therapy.
27. Current or treatment with another investigational drug within the previous 4 weeks.
28. Breast-feeding or pregnant women, no effective contraception if risk of conception exists (up to 4 months after end of chemotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Overall Survival (OS) at 18 months since randomization of patients with GBM treated in the experimental arm with UCPVax +/- pembrolizumab combined with standard treatment (Temozolomide +/- Novo-TTF-200A) | 18 months
  Rate for patients alive at 18 months post-randomization

SECONDARY OUTCOMES:
Assessment of the Overall Survival (OS) at 18 months since randomization of patients with GBM treated in the control arm receiving standard treatment( Temozolomide +/- NovoTTF-200A) | 18 months
  The rate of patients alive at 18 months post randomization
Assessment of the Overall Survival (OS) in the three arms | from date of randomization until date of death from any cause, assessed up to 42 months
  Overall survival (OS) defined as the time interval from randomization to the date of death from any cause. Alive patients will be censored at the last date known to be alive, either during study treatment period or during follow-up period
Assessment of the progression free survival (PFS) since randomization in the three arms | From date of randomization until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 42 months
  Progression free survival (PFS) according to RANO 2.0 criteria: defined as the time interval from the date of randomization to the date of first documented disease progression or death from any cause, whichever occurs first. Alive patients without progression will be censored at last radiological evaluation showing no progression during study treatment follow-up.
Assessment of the progression free survival (PFS) at 6 months since randomization in the three arms | 6 months
  Progression free survival (PFS) according to RANO 2.0 criteria: defined as the time interval from the date of randomization to the date of first documented disease progression or death from any cause, whichever occurs first. Alive patients without progression will be censored at last radiological evaluation showing no progression during study treatment follow-up.
Evaluation of incidence of treatment-emergent adverse events in the three arms | up to 42 months
  Adverse events and routine lab abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), timing, seriousness and relationship to study treatments at each visit.
Assessment of the immunogenicity of the proposal combination therapy. | average of 30 months
  UCP specific TCD4 T-cell response will be assess by ex vivo IFN-γ ELISpot in peripheral blood (Adotevi JCO 2023).
Evaluation of health-related quality of life (HrQoL) in the two arms | up to 42 months
  Health related Quality of life will be evaluated with EORTC-QLQC30 questionnaire and BN20 module at randomization and at 6 months.
Exploratory biomarker study | average of 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier ADOTEVI, MD, Principal Investigator — University Hospital of Besançon; Antoine CARPENTIER, MD, Principal Investigator — University Hospital of Besançon
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - Centre Georges François Leclerc, Dijon
  - CHU La Timone, Marseille
  - Hôpital Saint-Louis - APHP, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laheurte C, Boullerot L, Ndao B, Malfroy M, Queiroz L, Guillaume P, Loyon R, Seffar E, Gravelin E, Renaudin A, Jacquin M, Meurisse A, Vernerey D, Ghiringhelli F, Godet Y, Genolet R, Jandus C, Borg C, Adotevi O. UCPVax, a CD4 helper peptide vaccine, induces polyfunctional Th1 cells, antibody response, and epitope spreading to improve antitumor immunity. Cell Rep Med. 2025 Jul 15;6(7):102196. doi: 10.1016/j.xcrm.2025.102196. Epub 2025 Jun 20. PMID 40543509
- [Background] Adotevi O, Vernerey D, Jacoulet P, Meurisse A, Laheurte C, Almotlak H, Jacquin M, Kaulek V, Boullerot L, Malfroy M, Orillard E, Eberst G, Lagrange A, Favier L, Gainet-Brun M, Doucet L, Teixeira L, Ghrieb Z, Clairet AL, Guillaume Y, Kroemer M, Hocquet D, Moltenis M, Limat S, Quoix E, Mascaux C, Debieuvre D, Fagnoni-Legat C, Borg C, Westeel V. Safety, Immunogenicity, and 1-Year Efficacy of Universal Cancer Peptide-Based Vaccine in Patients With Refractory Advanced Non-Small-Cell Lung Cancer: A Phase Ib/Phase IIa De-Escalation Study. J Clin Oncol. 2023 Jan 10;41(2):373-384. doi: 10.1200/JCO.22.00096. Epub 2022 Sep 7. PMID 36070539